CLINICAL TRIAL: NCT02521415
Title: Randomized Controlled Trial of Intranasal Ketamine Compared to Intranasal Fentanyl for Analgesia in Children With Suspected, Isolated Extremity Fractures in the Pediatric Emergency Department
Brief Title: IN Sub-Dissociative Ketamine vs IN Fentanyl
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Carolinas Trauma Network Research Group (Unknown); Charlotte, Houston, Milwaukee Prehospital Emergency Research Nodal Center-CHaMP-ERNC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INK-2015
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2018-02

CONDITIONS: Bone Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Ketamine; Fentanyl; Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine (Experimental): ketamine (1mg/kg)
  Interventions: Drug: ketamine; Drug: ibuprofen or acetaminophen
- fentanyl (Active Comparator): fentanyl (1.5 micrograms/kg)
  Interventions: Drug: fentanyl; Drug: ibuprofen or acetaminophen

INTERVENTIONS:
Drug: ketamine — intranasal (IN) sub-dissociative ketamine (1mg/kg)
  Other Names: intranasal pain medication
  Arms: ketamine
Drug: fentanyl — Intranasal (IN) fentanyl (1.5 micrograms/kg)
  Other Names: intranasal pain medication
  Arms: fentanyl
Drug: ibuprofen or acetaminophen — 10 mg/kg of ibuprofen or 15 mg/kg of acetaminophen will be given to participants prior to the randomized intervention

SUMMARY:
This single center, randomized control, double blind trial will prospectively examine the feasibility of intranasal, sub-dissociative (IN) ketamine versus intranasal fentanyl for pain control in the pediatric emergency department setting. The investigators hypothesize that IN ketamine may provide a safe and effective alternative to IN fentanyl for children with suspected, isolated extremity fractures.

Eighty children ages 3-17 years with a suspected, isolated extremity fracture that requires analgesia will be randomized to receive IN ketamine or IN fentanyl upon presentation to the emergency department and will be followed for 2 hours for efficacy and 6 hours for safety.

DETAILED DESCRIPTION:
Intranasal medications are commonly used in place of parenteral opioids in children. IN fentanyl is the most commonly used intranasal analgesic medication in the pediatric population with demonstrated safety and efficacy comparable to IV fentanyl and IV morphine. IN ketamine, at sub-dissociative doses, offers similar safety and efficacy to IN fentanyl and the additional advantage of potentially reducing the total use of opioid agents during the emergency department visit. Ketamine is easily stored and has a wide therapeutic window with an extremely low risk of cardiorespiratory complications. This study will compare the safety and efficacy of IN ketamine to IN fentanyl in children with suspected, isolated extremity fractures in the pediatric emergency department.

The primary aim of the study is to examine the feasibility of future protocol expansion. The investigators will conclude that additional studies are NOT feasible if the observed rate of side effects for ketamine that exceeds fentanyl by three-fold or event rate of 5% or more for ketamine-related SAEs. The primary aim of the study will compare the frequency of adverse events over 6-hours among children randomized to receive either intranasal sub-dissociative ketamine (IN ketamine) or intranasal fentanyl (IN fentanyl) for pain control in the emergency department. The exploratory aim of the study will compare the efficacy of intranasal ketamine to intranasal fentanyl as measured by a reduction in age appropriate pain scale scores over 2-hours. The secondary aim of the study will compare the total dose of opioid pain medication in morphine equivalents/kg/hour required during the ED evaluation of children with suspected, isolated extremity fractures after randomization and treatment with IN ketamine or IN fentanyl.

Eighty children ages 3-17 years with a suspected, isolated extremity fracture that requires analgesia will be randomized to receive IN ketamine or IN fentanyl upon presentation to the emergency department and will be followed for 2 hours for efficacy and 6 hours for safety.

All participants will be premedicated with acetaminophen or ibuprofen and baseline data, including pain level, will be collected. The trial consists of two treatment arms. (IN ketamine 1 mg/kg or IN fentanyl 1.5 mcg/kg). Randomization will follow a 1:1 ratio, with approximately 40 per group. Randomization will be stratified by ages 3-10 and 11-17. The participants will be assessed by a research coordinator for adverse events every 5 minutes using an adverse events checklist for the first fifteen minutes post study medication administration and every 30 minutes for the first two hours after drug administration. The vital signs and pain scale assessment will be repeated every 10 minutes for the first 30 minutes and then every 30 minutes for the first two hours after drug administration. A final assessment will be made 6 hours after the last dose of study drug or at discharge from the ED to assess for late side effects or adverse events. Study medication may be repeated times one at a reduced dose after 20 minutes when the full effects of the first dose are known. The decision to administer additional study medication (0.5 mg/kg ketamine or 0.75 mcg/kg fentanyl ) will at be at the discretion of the treating physician. Should a second dose of study medication be required, a new schedule of patient assessments will commence following the same schedule as for the first dose. Participant assessments will continue until the 2 hour endpoint is reached from the time of the last drug administration, with a final assessment at 6 hours after the last dose of study drug or at discharge from the ED to assess for late side effects or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* single suspected, isolated extremity fracture that requires analgesia

Exclusion Criteria:

* GCS < 15 at ED presentation,
* reported allergy or adverse reaction to ketamine or fentanyl,
* pregnancy,
* intoxication,
* hypotension (less than 70 mmHg +2x age or less than 90 mm Hg for patients greater than 11 years of age)
* weight > 70 kg
* patients receiving opioid analgesia administered prior to arrival
* multiply injured patients (injuries to multiple extremities)
* aberrant nasal anatomy that precludes IN medications

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Reynolds, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center Main - Levine Children's Hospital Emergency Department, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Reynolds SL, Studnek JR, Bryant K, VanderHave K, Grossman E, Moore CG, Young J, Hogg M, Runyon MS. Study protocol of a randomised controlled trial of intranasal ketamine compared with intranasal fentanyl for analgesia in children with suspected, isolated extremity fractures in the paediatric emergency department. BMJ Open. 2016 Sep 8;6(9):e012190. doi: 10.1136/bmjopen-2016-012190. PMID 27609854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Fentanyl
Started | 43 | 44
Completed | 43 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: pain score at baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Fentanyl | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Customized [Count of Participants; unit: Participants]
  4-10 years | 30 | 32 | 62
  11-17 years | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 26 | 28 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/black | 10 | 8 | 18
  White | 22 | 26 | 48
  American Indian/Alaskan native | 1 | 0 | 1
  Other | 10 | 10 | 20
  Hispanic or Latino | 7 | 12 | 19
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome: Number of Participants With Minor Side Effects and Significant Adverse Events
Description: We will conclude that such a study is NOT feasible if we observe a rate of side effects for ketamine that exceeds fentanyl by three-fold or event rate of 5% or more for ketamine-related significant adverse events. Side effects are common events experienced by patients receiving ketamine or fentanyl that do not change outcomes for the patient but may affect the patient experience. A significant adverse event (SAE) includes any adverse event that begins after the short form consent has been completed that causes a threat to life, limb or an organ system, causes prolongation of hospitalization, or requires new medical or surgical treatment to correct.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 43 | 44
Participants
  serious adverse events | 0 | 0
  non-serious adverse events | 41 | 25
  no AEs observed | 2 | 19

2. Secondary Outcome: Secondary Outcome: Total Dose of Opioid Pain Medication in Morphine Equivalents/kg/Hour
Description: Compare the total dose of opioid pain medication in morphine equivalents/kg/hour required during the ED evaluation of children with suspected forearm fractures after randomization and treatment with IN ketamine or IN fentanyl.
Time Frame: participants will be followed during the emergency department length of stay, estimated to average 6 hours
Measure: Median (Inter-Quartile Range); unit: morphine equivalents/kg/hr
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 43 | 44
morphine equivalents/kg/hr | 0.04 [0.02 to 0.11] | 0.05 [0.04 to 0.08]

3. Other Pre Specified Outcome: Exploratory Outcome: Reduction in Age Appropriate Pain Scale Scores
Description: Mean difference in the reduction of the pain scale scores at 20 minutes. Two commonly used, age appropriate and previously validated, pediatric pain assessment tools were used: FACES Pain Scale - Revised for children ages 4-10 and the Visual Analog Scale for children ages 11-17. The FACES Pain Scale - Revised is a self-reported measure of pain intensity developed for children with pain intensity represented by images of grimacing faces on a scale of 0 (no pain) to 10 (maximum pain). The Visual Analog Scale is a self-reported measure of pain intensity where patients mark their pain level on a 10 cm line that represents a continuum of no pain at 0 cm and worst pain at 10 cm. For analysis, pain scale data were merged and reported as values form 0 to 100. The minimum clinically significant reduction in pain was defined as a decrease of 20.
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 43 | 44
units on a scale | 44 (36) | 35 (29)

4. Other Pre Specified Outcome: Secondary Safety Outcome: Adverse Events Over 6 Hours
Description: Compare the frequency of types of adverse events over 6-hours among children randomized to receive either intranasal sub-dissociative ketamine (IN ketamine) or intranasal fentanyl (IN fentanyl) for pain control in the emergency department.
Time Frame: 6 hours
Population: Data were collected but all secondary outcomes for the study have not yet been analyzed
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Hour 6
Arm/Group | Ketamine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 41/43 | 25/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=43) | Fentanyl (N=44)
any adverse event (General disorders) | 41 (41) | 25 (25)
bad taste in mouth/throat (General disorders) | 37 (37) | 9 (9)
dizziness (Nervous system disorders) | 30 (30) | 6 (6)
sleepiness (General disorders) | 19 (19) | 15 (15) — includes patient reports of sleepiness, tiredness, or increased sleepiness among patients who were observed to be wide awake and conversant
drowsiness (General disorders) | 6 (6) | 3 (3)
itchy nose (General disorders) | 10 (10) | 9 (9)
visual disturbance (Eye disorders) | 4 (4) | 1 (1) — includes patient report of blurry vision, fuzzy vision, seeing a blue spot and seeing multiples
dysphoria (General disorders) | 1 (1) | 2 (2)
nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes